CLINICAL TRIAL: NCT05178303
Title: Composition for Treating Cirrhosis and Liver Cancer
Brief Title: Composition for Treating Cirrhosis and Liver Cancer (SB-1121)
Acronym: SB-1121
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nguyen Thi Trieu, MD (Individual)
Collaborators: Tran Minh Duc (Unknown)
Responsible Party: Sponsor-Investigator, Nguyen Thi Trieu, MD, Scientific Manager, Trieu, Nguyen Thi, M.D.
Organization: Trieu, Nguyen Thi, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cirrhosis and Hcc
Expanded Access: NCT01198860 (Approved for marketing)
Record Dates: First submitted 2021-12-01; First posted 2022-01-05 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cirrhosis of the Liver
Keywords: Liver; Cirrhosis; Hcc; Flavonoids; Pregnenolone; Ascorbic acid; B6
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cirrhosis (Experimental): Experimental benefits in resistance to cirrhosis were observed in all patients who had previously received certain components of the treatment for cirrhosis SB-1121(1) for various therapeutic purposes.
  Interventions: Drug: SB-1121(1)
- Cirrhosis/Hcc "stable" (Experimental): Experimental benefits in resistance to cirrhosis/Hcc were observed in all patients who had previously received certain components of the treatment for cirrhosis SB-1121(2) for various therapeutic purposes.
  Interventions: Drug: SB-1121(2)

INTERVENTIONS:
Drug: SB-1121(1) — The daily maintenance, SB-1121(1) dose is to take 2 times a day, 1 tablet each time.
  Other Names: Cirrhosis/SB-1121
  Arms: Cirrhosis
Drug: SB-1121(2) — The daily maintenance, SB-1121(2) dose is to take 2 times a day, 1 tablet each time.
  Other Names: Cirrhosis/Hcc/SB-1121
  Arms: Cirrhosis/Hcc "stable"

SUMMARY:
The composition treats cirrhosis and hepatocellular carcinoma (Hcc) at an early stage. The product is extracted from herbs, including Adenosma glutinosum extract, Eclipta prostrata extract, Phyllanthus urinaria extract, Impatiens balsamina extract, Ascorbic acid, pyridoxine 5-phosphate, L-Arginine hydrochloride, Pregnenolone acetate. These components have participated in repairing and regenerating new liver parenchyma, preventing fibrosis cell generation, preventing liver cancer cell growth at an early stage. The composition supplements precursors which help the body strengthen antibodies and reduce the risk of inflammation, restore physiological and biochemical functions of liver cells after chronic inflammation.

DETAILED DESCRIPTION:
The composition is fractionally extracted from herbs. Flavonoids, isoflavonoids, and pregnenolone combined with ascorbic acid, pyridoxine 5-phosphate, L-arginine act as the key compounds in the regeneration of fibrosis liver cells, remove scar tissue, stimulate and release growth hormones, prevent progression to Hcc and prevent Hcc recurrence.

The pharmaceutical ingredients involved in the composition are calculated to increase their effectiveness in preventing and curing cirrhosis and Hcc.

Currently, many preparations have been and are being studied to fight against cirrhosis and liver cancer globally. The effectiveness of this preparation is a new finding which has been proven over 5 years of follow-up.

Pregnenolone is a cortisol precursor. Cortisol plays an important role in several systems in the body, including the immune system(in the cycle of the immune system to produce B lymphocytes). This ingredient is used as a supplement to stabilize the endothelium, regulate the amount of cortisol within normal limits, and help the body produce B lymphocytes with a good response.

Kaempferol is a flavonoid that participates in cell protection against toxic proteins which were produced during prolonged inflammation; blocking the action and removing denatured proteins that change the parenchyma of liver cells. The selected flavonoids repaired the fibrotic structure of liver parenchyma after chronic inflammation. Ascorbic acid, pyridoxine 5-phosphate, and L-arginine help to facilitate biological functions in cell adhesion, synergize with flavonoids in cell membrane protection, structural repair, and liver cell regeneration.

Ascorbic acid, pyridoxine 5-phosphate act as enzymes that catalyze processes conveniently.

ELIGIBILITY:
Inclusion Criteria:

* All patients with underlying medical conditions who have been taking medications for these conditions.
* Patients with AIDS, HIV, HBV, HCV, and patients with co-infections.
* The cancer patients are stable.
* Patients with congenital or acquired immunodeficiency.

Exclusion Criteria:

* Unstable cancer patients.
* Decompensated cirrhosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
The test uses sound waves to measure the stiffness of liver tissue on patient cirrhosis (Arm 1) | 36 months
  HBV, HCV,... injure healthy liver cells, causing cell death and inflammation. Healthy liver tissue is replaced with scar tissue and the liver is damaged.

SECONDARY OUTCOMES:
The test uses sound waves to measure the stiffness of liver tissue on patient cirrhosis/Hcc (Arm 2) | 36 months
  Hepatocellular carcinoma occurs most often in people with chronic liver diseases, cirrhosis, such as cirrhosis caused by hepatitis B, hepatitis C infection,...

CONTACTS AND LOCATIONS:
Overall Officials: Tran Minh Cam Tu, Dr., Principal Investigator — Saigon Biopharma Company Limited
Locations (2):
- Saigon Biopharma LLC, Wilmington, Delaware, United States
- Saigon Biopharma Company Limited, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Raza A, Sood GK. Hepatocellular carcinoma review: current treatment, and evidence-based medicine. World J Gastroenterol. 2014 Apr 21;20(15):4115-27. doi: 10.3748/wjg.v20.i15.4115. PMID 24764650
- [Result] Kalra A, Yetiskul E, Wehrle CJ, Tuma F. Physiology, Liver. 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK535438/ PMID 30571059
- [Result] Naran K, Nundalall T, Chetty S, Barth S. Principles of Immunotherapy: Implications for Treatment Strategies in Cancer and Infectious Diseases. Front Microbiol. 2018 Dec 21;9:3158. doi: 10.3389/fmicb.2018.03158. eCollection 2018. PMID 30622524
- [Result] Roth A, Schaffner W, Hertel C. Phytoestrogen kaempferol (3,4',5,7-tetrahydroxyflavone) protects PC12 and T47D cells from beta-amyloid-induced toxicity. J Neurosci Res. 1999 Aug 1;57(3):399-404. PMID 10412031
- [Result] Flisiak R. Role of Ito cells in the liver function. Pol J Pathol. 1997;48(3):139-45. PMID 9401406
- [Result] Kaestner KH. Progress in molecular biology and translational science. development, differentiation and disease of the para-alimentary tract. Preface. Prog Mol Biol Transl Sci. 2010;97:xi-xii. doi: 10.1016/B978-0-12-385233-5.00015-5. No abstract available. PMID 21074727
- [Result] 19. IPSC-derived 3D human fatty liver models Maddalena Parafati, Siobhan Malany, in iPSCs in Tissue Engineering, 2021
- [Result] Hennedige T, Venkatesh SK. Imaging of hepatocellular carcinoma: diagnosis, staging and treatment monitoring. Cancer Imaging. 2013 Feb 8;12(3):530-47. doi: 10.1102/1470-7330.2012.0044. PMID 23400006
- See also: Liver Cancer Risk Factors — http://www.cancer.org/cancer/liver-cancer/causes-risks-prevention/risk-factors.html
- See also: Viral Hepatitis and Liver Disease — http://www.hepatitis.va.gov/cirrhosis/background/stages.asp
- See also: What does the liver do — http://www.medicalnewstoday.com/articles/305075
- See also: Flavonoids as Multi-target Inhibitors for Proteins Associated with Ebola Virus: In Silico Discovery Using Virtual Screening and Molecular Docking Studies — http://pubmed.ncbi.nlm.nih.gov/26286008/
- See also: Vitamin C Is an Essential Factor on the Anti-viral Immune Responses through the Production of Interferon-α/β at the Initial Stage of Influenza A Virus (H3N2) Infection — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3659258/
- See also: The antiviral properties of vitamin C — http://pubmed.ncbi.nlm.nih.gov/31852327/